CLINICAL TRIAL: NCT02514031
Title: A Phase I/Ib, Single-Arm, Open-Label, Multi-Center Trial Using ARQ-761 (Beta-Lapachone) Treatment With Gemcitabine/Nab-Paclitaxel Chemotherapy In Metastatic, Unresectable, Or Recurrent Pancreatic Cancer
Brief Title: ARQ-761 Treatment With Gemcitabine/Nab-Paclitaxel Chemotherapy In Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study placed on temporarily hold to enrollment due to quality testing necessary for the study drug.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Muhammad Beg, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STU 052015-024
Record Dates: First submitted 2015-06-17; First posted 2015-08-03 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — beta-lapachone; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARQ-761 (Experimental): A 2 week lead-in monotherapy of ARQ-761 (The amount of ARQ-761 that will be given to the participant will depend on the time at which the participant was enrolled in the study
  Afterwards the 28-day cycle of combination treatment of ARQ-761 along with gemcitabine (1000 mg/m2) + nab-paclitaxel (125 mg/m2) will begin.
  Interventions: Drug: ARQ-761; Drug: Gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: ARQ-761 — Dose Level 1:
  ARQ761 195 mg IV D1, D15 Gemcitabine 1000 mg/m2 D1, 8, 15 Nab paclitaxel 125 mg/m2 D1, 8, 15
  Dose Level 2:
  ARQ761 290 mg IV D1, D15 Gemcitabine 1000 mg/m2 D1,8,15
  Dose Level 3:
  ARQ761 390 mg IV D1, D15 Gemcitabine 1000 mg/m2 D1,8,15 Nab-paclitaxel 125 mg/m2 D1,8,15
  Expansion Dose Level:
  ARQ761 390 IV mg or as tolerated D1, 15 Gemcitabine 1000 mg/m2 D1,8,15 Nab-Paclitaxel 125 mg/m2 D1,8,15
  Other Names: Beta-Lapachone
Drug: Gemcitabine — Therapy after lead in Phase:
  You will receive Gemcitabine (1000mg/m2) administered intravenously on Days 1,8, 15-every 28 days. All cycles are 28 days in duration and there are no rest periods between cycles. You may continue treatment after cycle 6 until disease progression.
  Other Names: Gemzar
Drug: nab-paclitaxel — Therapy after lead in phase:
  You will receive nab-paclitaxel (125 mg/m2) administered intravenously on Days 1,8, 15-every 28 days. All cycles are 28 days in duration and there are no rest periods between cycles. You may continue treatment after cycle 6 until disease progression.
  Other Names: Abraxane

SUMMARY:
This is a study of ARQ-761 (beta-lapachone) with gemcitabine/nab-paclitaxel chemotherapy in subjects with advanced (metastatic, unresectable, or recurrent) pancreatic cancer that has not been treated with gemcitabine.

DETAILED DESCRIPTION:
Screening:

* Demographic information (age, gender, race, ethnic origin).
* Physical exam and review of your past and present medical history including any surgeries a and/or infections;
* Vital signs (temperature, pulse, respirations, blood pressure); height, weight;
* Concurrent medications (medications whether prescribed or over-the counter that you have taken or are currently taking);
* Performance Status (how well you are able to perform daily activities)
* Review of any side effects that you may have experienced or may be experiencing before receiving the study drug and medications
* Blood will be collected for routine lab tests
* Urinalysis
* Pregnancy Test (if you are a woman of child-bearing potential)
* Radiologic evaluation (review of any CT scans you may have had)
* Tumor measurements:
* A CT scan (chest/abdomen/pelvis) is a special test that produces an image of your body using a. small amount of radiation. The image shows the body tissues and structures in three dimensions (3-D).
* Electrocardiogram (EKG), a tracing of the electrical activity of the heart;
* Oxygen saturation (measures how much oxygen the blood is carrying)
* Biopsy for correlative studies - if archived tumor specimen cannot be obtained, you will need to undergo a fresh biopsy
* Completion of a Quality of life questionnaire

This visit may last approximately 1-2 hours. Visits that included radiologic evaluation may last longer, approximately 2-3 hours.

The treatment consists of:

* A 2 week lead-in monotherapy of ARQ-761 - they will receive the current dose of ARQ761 alone

  o The amount of ARQ-761 that will be given to you will depend on the time at which you are enrolled in the study.
* Afterwards the 28-day cycle of combination treatment of ARQ-761 along with gemcitabine (1000 mg/m2) + nab-paclitaxel (125 mg/m2) will begin

Lead-in 2 weeks before the combination therapy begins:

Monotherapy of ARQ-761

Day 1:

* Vital signs
* Review of medical history
* Physical exam
* Review of any medications they are taking or have taken
* Review of any adverse events they may have experienced
* Performance status evaluation (questions about their activity level)
* Quality of life assessment questionnaire
* Blood will be drawn for routine laboratory tests
* Urinalysis
* Oxygen saturation measurement using a finger light sensor
* EKG
* ARQ761 Administration via intravenous (IV) for approximately 120 minutes Clinic Visit: 3 - 3 ½ Hours

Combination Therapy:

Cycle 1 Day 1

* Vital signs
* Review of medical history and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Quality of life assessment questionnaire
* Blood work
* Blood for correlative studies
* Urinalysis
* EKG
* Oxygen saturation measurement using a finger light sensor

Combination Treatment regimen:

* Nab-Paclitaxel administered via intravenous (IV) over 30 minutes then;
* Gemcitabine administered via intravenous (IV) over 30 minutes

After waiting for 60 minutes (1 hour) then:

* ARQ 761 administered via intravenous (IV) over 120 minutes (2 hours)
* Biopsy of their tumor
* PKs (pharmacokinetics) (consist of drawing of approximately ½ teaspoon of blood to determine what their body does to the study drug) will be collected at:

  * Pre-Infusion of ARQ-761
  * 30 minutes after beginning of infusion
  * 1, 2, and 4 hour post-infusion of ARQ-761
* PDs (pharmacodynamics) (consist of drawing of approximately ½ teaspoon of blood to examine the response of protein biomarkers in patients treated with ARQ-761during the clinical trial) will be collected:

  * Pre-infusion of ARQ-761
  * 3 hour post-infusion of ARQ-761

Clinic Visit: 8 Hours

Cycle 1 Day 8

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Blood work
* Nab-Paclitaxel administered via intravenous (IV) over 30 minutes then;
* Gemcitabine administered via intravenous (IV) over 30 minutes

Clinic Visit: 2 hours

Cycle 1 Day 15

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Blood work
* Blood for correlative studies
* Urinalysis
* EKG
* Oxygen saturation measurement using a finger light sensor

Treatment regimen:

* Nab-Paclitaxel administered via intravenous (IV) over 30 minutes then;
* Gemcitabine administered via intravenous (IV) over 30 minutes

After waiting for 60 minutes (1 hour) then:

* ARQ 761 administered via intravenous (IV) over 120 minutes (2 hours)
* PKs (pharmacokinetics) (consist of drawing of approximately ½ teaspoon of blood to determine what their body does to the study drug) will be collected at:

  * Pre-Infusion of ARQ-761
  * 30 minutes after beginning of infusion
  * 1, 2, and 4 hour post-infusion of ARQ-761
* PDs (pharmacodynamics) (consist of drawing of approximately ½ teaspoon of blood to examine the response of protein biomarkers in patients treated with ARQ-761during the clinical trial) will be collected:

  * Pre-infusion of ARQ-761
  * 3 hour post-infusion of ARQ-761

Clinic Visit: 8 hours

Cycle 2 Day 1

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Oxygen saturation measurement using a finger light sensor
* Blood work
* Urinalysis
* Oxygen saturation measurement using a finger light sensor
* Quality of life assessment

Combination treatment regimen same as for Cycle 1 Day 1

Clinic Visit: 5 - 6 hours

Cycle 2 Day 8

* Vital signs
* A nurse will ask them general screening questions
* Blood work
* Nab-Paclitaxel administered via intravenous (IV) over 30 minutes then;
* Gemcitabine administered via intravenous (IV) over 30 minutes

Clinic Visit: 2-3 hours

Cycle 2 Day 15

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Blood work
* Urinalysis
* Oxygen saturation measurement using a finger light sensor

Combination treatment regimen same as for Cycle 1 Day 1

Clinic Visit: 5 - 6 hours

Cycle 2 Day 27

• CT scan of their chest/abdomen/pelvis

Clinic Visit: 1 - 2 hours

Cycle 3 and all subsequent odd cycles Day 1

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Quality of life assessment questionnaire
* Blood work
* Urinalysis
* Oxygen saturation measurement using a finger light sensor

Combination treatment regimen same as for Cycle 1 Day 1

Clinic Visit: 5 - 6 hours

Cycle 3 and all subsequent odd cycles Day 8

* Vital signs
* A nurse will ask them general screening questions
* Blood work
* Nab-Paclitaxel administered via intravenous (IV) over 30 minutes then;
* Gemcitabine administered via intravenous (IV) over 30 minutes

Clinic Visit: 2-3 hours

Cycle 3 and all subsequent odd cycles Day 15

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Blood work
* Urinalysis
* Oxygen saturation measurement using a finger light sensor
* Combination treatment regimen same as for Cycle 1 Day 1

Clinic Visit: 6 hours

Cycle 4 and all subsequent even cycles Day 1

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Quality of life assessment questionnaire
* Blood work
* Urinalysis
* Oxygen saturation measurement using a finger light sensor

Combination treatment regimen same as for Cycle 1 Day 1

Clinic Visit: 6 hours

Cycle 4 and all subsequent even cycles Day 8

* Vital signs
* A nurse will ask them general screening questions
* Blood work
* Nab-Paclitaxel administered via intravenous (IV) over 30 minutes then;
* Gemcitabine administered via intravenous (IV) over 30 minutes

Clinic Visit: 2-3 hours

Cycle 4 and all subsequent even cycles Day 15

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Blood work
* Urinalysis
* Oxygen saturation measurement using a finger light sensor

Combination treatment regimen same as for Cycle 1 Day 1

Clinic Visit: 6 hours

Cycle 4 and all subsequent even cycles Day 27

• CT scan of their chest/abdomen/pelvis

Clinic Visit: 1 - 2 hours

Off-Treatment Visit/End of Study Visit

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Quality of life assessment questionnaire
* Blood work
* Blood for correlative studies
* Urinalysis
* Oxygen saturation measurement using a finger light sensor

Clinic Visit: 1 - 2 hours

Follow-up Procedures

They will be seen once at 4 weeks after completion of (or early withdrawal from) study treatment. This visit will be repeated every 4 weeks until resolution of any side effects. The following will be done at this visit:

* Vital signs
* History and physical exam
* Performance status evaluation (questions about their activity level)
* Toxicity evaluation (questions about their side effects)
* Blood work

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically or cytologically confirmed pancreatic adenocarcinoma that is metastatic, unresectable, or recurrent.
2. Has received at most 1 line of prior non-gemcitabine chemotherapy for:

   * metastatic/unresectable disease.
   * Prior adjuvant gemcitabine, if completed more than 12 months prior to enrollment is not considered as prior line of therapy.
   * Radiosensitizing chemotherapy will not be considered a prior line of therapy.
3. Prior and concurrent therapy4. Measurable disease is required per RECIST criteria 1.1.

5. Age ≥18 years. 6. ECOG performance status 0 or 1 7. Anticipated life expectancy ≥ three months. 8. Central venous access 9. Availability of unstained slides or paraffin block tissue from archived tumor specimen. If not available the subject will undergo a fresh biopsy.

10. Specific pretreatment clinical laboratory parameters that are required within 14 days prior to registration.

11. Subjects must be recovered from any toxicity related to prior anti-neoplastic therapy (to grade <1).

12. Women of child-bearing potential and men must agree to use adequate contraception hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria:

1. Receiving any other investigational agents.
2. Subjects with known untreated brain metastases.
3. Subjects receiving hepatic enzyme-inducing antiseizure drugs ("EIASD
4. Uncontrolled intercurrent illness
5. Pregnancy
6. Any significant medical condition, laboratory abnormality, or psychiatric illness. 7. Any condition including the presence of laboratory abnormalities.

8. Any condition that confounds the ability to interpret data from the study. 9. Unwillingness or inability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Day 8, Day 1 and Day 15 every 28 days for 168 days or until disease progression, Off Treatment (Up to 8 months) , and 4 weeks after treatment.
  Determine the maximum tolerated dose (MTD) of ARQ761 when given in combination with gemcitabine and nab-paclitaxel (GEM-Nab-Pac).

SECONDARY OUTCOMES:
Safety will be assessed by quantifying toxicities using the NCI's CTCAE v4.0 toxicity criteria | Day 8 , Day 1 and Day 15 every 28 days for 168 days or until disease progression, Off Treatment (Up to 8 months) , and 4 weeks after treatment.
  Safety will be assessed by quantifying toxicities using the NCI's CTCAE v4.0 toxicity criteria.
Overall Response Rate | Imaging will be done every 2-3 months until you are off treatment (Up to 8 months).
  CT Chest/Abdomen/Pelvis to determine clinical activity as defined by overall response rate (ORR).
Progression Free Survival | Imaging will be done every 2nd cycle starting with week 10 (cycle 2) until you are off treatment (Up to 8 months).
  CT Chest/Abdomen/Pelvis to determine clinical activity as defined by Progression Free Survival .
Time To Progression | Imaging will be done every 2nd cycle starting with week 10 (cycle 2) until you are off treatment (Up to 8 months).
  CT Chest/Abdomen/Pelvis to determine clinical activity as defined by Time To Progression.
Pharmacokinetic Profile | During Cycle 1 Day 1 and Cycle 1 Day 15
  The pharmacokinetic profile of ARQ761 will be determined by measurement of blood levels at predetermined time points.
Tolerability | Day 8, Day 1 and Day 15 every 28 days for 168 days or until disease progression, Off Treatment (Up to 8 months) , and 4 weeks after treatment.
  Tolerability will be assessed by quantifying toxicities using the NCI's CTCAE v4.0 toxicity criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Beg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - UT Southwestern Medical Center, Dallas, Texas